CLINICAL TRIAL: NCT05191771
Title: Multicentric, Randomized, Comparative Clinical Study on the Evaluation of the Efficacy and Safety of Neovis® Total Multi Versus Systane® Balance on the Treatment of Ocular Dryness Associated With Meibomian Gland Dysfunction
Brief Title: Evaluation of Neovis® Total Multi Versus Systane® Balance on Ocular Dryness Associated With Meibomian Gland Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Horus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21E1007
Record Dates: First submitted 2021-12-10; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational product (Experimental)
  Interventions: Device: Neovis Total Multi
- Comparator (Active Comparator)
  Interventions: Device: Systane Balance

INTERVENTIONS:
Device: Neovis Total Multi — 1 drop in each eye, 4 times per day
  Arms: Investigational product
Device: Systane Balance — 1 drop in each eye, 4 times per day
  Arms: Comparator

SUMMARY:
This study is a multicentric, comparative, randomized, investigator-blinded, in parallel groups study to demonstrate the non-inferiority of Neovis® Total Multi in comparison with Systane® Balance, in terms of improvement of stability of Tear film in patients with eye dryness associated to meibomian gland dysfunction, after 28 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presenting dry eye symptoms for at least 6 months.
* OSDI (Ocular Surface Disease Index) ≥ 18
* At least one eye eligible with:

  * sum of peripheral corneal and conjunctival staining ≥ 4 and ≤ 9 (Oxford 0-15 grading scheme) AND
  * sum of 3 measurements of Tear film Break-Up Time (TBUT) ≤ 15s
* Meibomian Gland Dysfunction on at least one eye (same eye eligible) with a score of 1 or higher for meibum quality score (from 0: clear to 3: toothpaste/obstruction) and evidence of partial or whole missing Meibomian Glands.
* Ability and willingness to apply eyelid hygiene during the whole study, including wash-out period.
* Having given freely and expressly his/her informed consent.
* Able to comply with the study requirements, as defined in the present CIP, at the Investigator's appreciation.
* In France: subject being affiliated to a health social security system.
* Female subjects of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after the study end.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject deprived of freedom by administrative or legal decision.
* Subject in a social or health institution
* Subject who is under guardianship or who is not able to express his/her consent.
* Use of contact lenses in either eye during the study.
* Far best-corrected visual acuity ≤ 1/10.
* Subject with severe ocular dryness with one of these conditions:

  * Eyelid or blinking malfunction
  * Corneal disorders not related to dry eye syndrome
  * Ocular metaplasia
  * Filamentous keratitis
  * Corneal neovascularization
* History of ocular traumatism, ocular infection or ocular inflammation within the last 3 months.
* History of ocular allergy or ocular herpes within the last 12 months.
* Subjects who underwent ocular surgery, including laser surgery, in either eye within the last 6 months.
* Any troubles of the ocular surface not related to dry eye syndrome.
* Use of the following ocular treatments: isotretinoïd, cyclosporine, tacrolimus, sirolimus, pimecrolimus during the month preceding the inclusion.
* IOP > 21 mmHg
* Uncontrolled systemic disease
* Alcohol abuse
* Psychiatric disorders
* Cognitive impairment that could affect evaluation of preferences or inability to understand written patient information
* Participation in other clinical studies in the last month
* Hypersensitivity to one or more components of the study product
* Dry eye due to systemic disease, concomitant medication, malign conditions or idiopathic causes
* Punctual plugs during the past 3 months
* Use of lipid-containing eye drops during the past 3 months
* Use of other therapeutic ophthalmics during the past 3 months
* Earlier participation at this clinical trial or the patient being an investigator or a member of the personnel involved at this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Tear-Film Break Up Time (TBUT) | 28 days
  Evaluation of the non-inferiority of Neovis® Total Multi in comparison with Systane® Balance, in terms of TBUT improvement, on worse eye

SECONDARY OUTCOMES:
Tear-Film Break Up Time (TBUT) (performance) | 84 days
  Main change from baseline of Tear-Film Break Up Time (TBUT) in the worse eye and contralateral eye
Cornea and conjunctiva staining (Oxford score) (performance) | 28 days
  Main change from baseline of cornea and conjunctiva staining (Oxford score) in the worse eye and contralateral eye
Cornea and conjunctiva staining (Oxford score) (performance) | 84 days
  Main change from baseline of cornea and conjunctiva staining (Oxford score) in the worse eye and contralateral eye
Meibomian gland expression (performance) | 28 days
  Main change from baseline of meibomian gland expression score in the worse eye and contralateral eye
Meibomian gland expression (performance) | 84 days
  Main change from baseline of meibomian gland expression score in the worse eye and contralateral eye
Meibum quality (performance) | 28 days
  Main change from baseline of meibum quality score in the worse eye and contralateral eye
Meibum quality (performance) | 84 days
  Main change from baseline of meibum quality score in the worse eye and contralateral eye
Meiboscopy (performance) | 28 days
  Main change from baseline of the number of partially missing or dropout meibomian glands in the worse eye and contralateral eye
Meiboscopy (performance) | 84 days
  Main change from baseline of the number of partially missing or dropout meibomian glands in the worse eye and contralateral eye
Eyelid margin abnormalities (performance) | 28 days
  Main change from baseline of the eyelid margin abnormalities score in the worse eye and contralateral eye
Eyelid margin abnormalities (performance) | 84 days
  Main change from baseline of the eyelid margin abnormalities score in the worse eye and contralateral eye
OSDI (questionnaire) (performance) | 28 days
  Main change from baseline of OSDI (Ocular Surface Disease Index) in the worse eye and contralateral eye
OSDI (questionnaire) (performance) | 84 days
  Main change from baseline of OSDI (Ocular Surface Disease Index) in the worse eye and contralateral eye
Global performance by the investigator (performance) | 28 days
  Global performance assessment by the investigator using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global performance by the investigator (performance) | 84 days
  Global performance assessment by the investigator using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global performance by the patient (performance) | 28 days
  Global performance assessment by the patient using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global performance by the patient (performance) | 84 days
  Global performance assessment by the patient using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global tolerance by the investigator (safety) | 28 days
  Global tolerance assessment by the investigator using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global tolerance by the investigator (safety) | 84 days
  Global tolerance assessment by the investigator using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global tolerance by the patient (safety) | 28 days
  Global tolerance assessment by the patient using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global tolerance by the patient (safety) | 84 days
  Global tolerance assessment by the patient using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Intensity of ocular symptoms upon instillation (safety) | 28 days
  Evaluation of intensity of ocular symptoms upon instillation on a scale from 0 (none) to 3 (severe)
Intensity of ocular symptoms upon instillation (safety) | 84 days
  Evaluation of intensity of ocular symptoms upon instillation on a scale from 0 (none) to 3 (severe)
Duration of ocular symptoms upon instillation (safety) | 28 days
  Evaluation of duration of ocular symptoms upon instillation in seconds/minutes/hours
Duration of ocular symptoms upon instillation (safety) | 84 days
  Evaluation of duration of ocular symptoms upon instillation in seconds/minutes/hours
Frequency of ocular symptoms upon instillation (safety) | 28 days
  Evaluation of frequency of ocular symptoms upon instillation on a scale from 1 (rarely) to 4 (very often)
Frequency of ocular symptoms upon instillation (safety) | 84 days
  Evaluation of frequency of ocular symptoms upon instillation on a scale from 1 (rarely) to 4 (very often)
Number of Adverse Events | 84 days
  Collection of ocular and systemic adverse events

OTHER OUTCOMES:
Non-Invasive Tear film Break-Up Time (NIBUT) (exploratory, optional) | 28 days
  Main change from baseline of Non-Invasive Tear film Break-Up Time (NIBUT) in the worse eye and contralateral eye
Non-Invasive Tear film Break-Up Time (NIBUT) (exploratory, optional) | 84 days
  Main change from baseline of Non-Invasive Tear film Break-Up Time (NIBUT) in the worse eye and contralateral eye
Lipid layer thickness (exploratory, optional) | 28 days
  Main change from baseline of lipid layer thickness with interferometry methods in the worse eye and contralateral eye
Lipid layer thickness (exploratory, optional) | 84 days
  Main change from baseline of lipid layer thickness with interferometry methods in the worse eye and contralateral eye
Functional visual acuity (exploratory, optional) | 28 days
  Main change from baseline of functional visual acuity in the worse eye and contralateral eye
Functional visual acuity (exploratory, optional) | 84 days
  Main change from baseline of functional visual acuity in the worse eye and contralateral eye
Super Oxyde Dismutase (SOD) dosage (exploratory, optional) | 84 days
  Main change from baseline of SOD1 and SOD2 in the worse eye
Goblet cells analysis (exploratory, optional) | 84 days
  Main change from baseline of Goblet cells in the worse eye

CONTACTS AND LOCATIONS:
Overall Officials: Hoffart Louis, Principal Investigator — Vision Sud

IPD SHARING:
Plan to Share IPD: Undecided
Depending on any journal publication of the results